CLINICAL TRIAL: NCT04185285
Title: Percutaneous Coronary Intervention Registry FRIBOURG
Acronym: Cardio-FR
Status: Recruiting | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Stéphane Cook, Prof, Chairman, cardiology, University of Freiburg
Other Study IDs: 003-REP-CER-FR-2
Record Dates: First submitted 2019-11-14; First posted 2019-12-04 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: PCI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous coronary intervention, stents

SUMMARY:
The registry aims to follow clinically all consecutive patients treated by percutaneous coronary interventions at hospital & university Fribourg.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients treated by percutaneous coronary intervention at our institution
* Able to give informed consent and willing to participate

Exclusion Criteria:

* Unwillingness to participate
* Enable to provide inform consent

Ages: 17 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient-oriented composite endpoints (POCE) | 2 years
  Academic Research Consortium definition
Major Bleeding | 2 years
  Bleeding Academic Research Consortium definition
Patient-oriented composite endpoints (POCE) | 5 years
  Academic Research Consortium definition
Major Bleeding | 5 years
  Bleeding Academic Research Consortium definition
Patient-oriented composite endpoints (POCE) | 10 years
  Academic Research Consortium definition
Major Bleeding | 10 years
  Bleeding Academic Research Consortium definition

SECONDARY OUTCOMES:
all-cause death | 2 years
  Academic Research Consortium definition
any revascularization | 2 years
  Academic Research Consortium definition
any myocardial infarction | 2 years
  Academic Research Consortium definition

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology, university Fribourg Medical Center, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cook ST, Allemann L, Cook M, Arroyo DA, Pittet T, Meier P, Togni M, Brahim-Mathiron A, Puricel S, Cook S. Sex differences in ST-segment elevation myocardial infarction patients treated by primary percutaneous intervention. Open Heart. 2025 Jan 4;12(1):e002831. doi: 10.1136/openhrt-2024-002831. PMID 39756819